CLINICAL TRIAL: NCT05008107
Title: Virtual Reality as a Perioperative Teaching Tool for Families: A Randomized Controlled Trial
Brief Title: Virtual Reality as a Perioperative Teaching Tool for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Brittany Willer, Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001402
Record Dates: First submitted 2021-07-26; First posted 2021-08-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Surgical Procedure, Unspecified; Tonsil Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual reality (VR) will be provided to families of patients undergoing ambulatory pediatric surgery. VR will provide personalized education to patients and their families about the entire continuum of the child's surgical experience. This will range from the hospital registration, the peri-operative experience, including the separation of the child from the parent in the pre-operative area and the anesthetic induction process, and the post-operative hospital ward.
  Interventions: Other: Virtual reality
- Control (No Intervention): Families will receive standard pre-operative instructions.

INTERVENTIONS:
Other: Virtual reality — Using VR goggles to watch peri-operative instructional video.
  Other Names: VR
  Arms: Virtual Reality

SUMMARY:
Commonly, families and providers have turned to internet-based resources to provide insight as to the perioperative experience. Though there is a large amount of information that is available on the internet, medical information on the internet is of highly variable quality and the information may be conflicting or inaccurate. It is hard for even the savvy well-educated patient and family to navigate and sift through all the information available. Therefore, generic web-based information does not necessarily decrease patient and caregiver anxiety. As an alternative, the investigators propose an interactive teaching tool utilizing virtual reality that may provide a cost-efficient, content-rich supplement to the traditional phone or internet-based patient education. Virtual reality (VR) will be provided to families of patients undergoing ambulatory pediatric surgery. VR will provide personalized education to patients and their families about the entire continuum of the child's surgical experience. This will range from the hospital registration, the peri-operative experience, including the separation of the child from the parent in the pre-operative area and the anesthetic induction process, and the post-operative hospital ward. The virtual reality (VR) tool will also review the in-hospital post-operative recovery process. The patient will be shown this either via an oculus headset or using their own smartphone device. In addition to improving a parent's comprehension of what their child will experience, the investigators expect that the virtual reality tool may also improve patient and caregiver satisfaction with the overall perioperative experience.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing tonsillectomy/adenotonsillectomy ± ear tubes in the ambulatory setting

Exclusion Criteria:

* Non-English speaking (VR program is currently only offered in English)
* Inpatient
* Unable to effectively use VR (blind, severe motion sickness)
* History of procedure in the operating room within the past year
* Having a combination/additional procedure

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Patient Pre-op Anxiety Score | Baseline
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Parent Pre-op Anxiety Score | Baseline
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Patient Post-op Anxiety Score | Immediately prior to discharge
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Parent Post-op Anxiety Score | Immediately prior to discharge
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
Parent Satisfaction Score | Immediately prior to discharge
  Assessed using an adaptation of the English version of the Leiden Perioperative Patient Satisfaction questionnaire (LPPSq). This questionnaire assesses 4 domains of satisfaction: information provision, professional competence, patient-staff relationship, and service with a total of 24 questions. Questions will be scored on a 1-5 Likert scale (from completely dissatisfied to completely satisfied) with the total satisfaction score ranging from 24-120 possible points.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States